CLINICAL TRIAL: NCT05904925
Title: Pilates Exercises for the Prevention of Musculoskeletal Complaints During Pregnancy: a Protocol of a Pilot Randomized Controlled Trial With Economic Evaluation
Brief Title: Pilates for the Prevention of Musculoskeletal Complaints During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Cristina Maria Nunes Cabral, Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 59486822.3.0000.8084
Record Dates: First submitted 2023-05-18; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pregnancy
Keywords: Pilates; Pregnancy; Randomized controlled trial; Pilot study; Musculoskeletal complaint; Economic evaluation
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Usual care group will perform the usual prenatal care indicated by the obstetrician and will receive an educational booklet.
- Pilates (Active Comparator): Pilates group will perform the usual prenatal care indicated by the obstetrician and will receive an educational booklet. Additionally, this group will receive an exercise program based on Pilates, twice a week, individually, throughout the gestational period.
  Interventions: Other: Pilates exercises

INTERVENTIONS:
Other: Pilates exercises — Sessions will last 60 minutes: five minutes for warming up, 50 minutes for the practice of Pilates exercises, and five minutes for relaxing with the Swiss ball. The exercise protocol will be divided into three gestational phases, covering the entire gestational period, with different and specific objectives for each phase. In all phases, the exercises will be classified into three levels of difficulty: basic, intermediate, and advanced, according to the evolution of each pregnant woman throughout the practice of Pilates. Modifications will be allowed to facilitate or hinder the execution of the movement. The exercises will be performed in one or two sets of seven to 10 repetitions. The number of series, repetitions and exercises and interval time between them, as well as the level of difficulty of the exercises, will be gradually adjusted. The intensity of the exercises will vary between light and moderate and will be controlled by the Borg scale.
  Arms: Pilates

SUMMARY:
The goal of this pilot randomized controlled trial with economic evaluation is to evaluate the viability of Pilates in the prevention of musculoskeletal complaints, throughout the entire gestational period, in pregnant women. The main question it aims to answer is if it is feasible to perform exercises during the entire gestational period to prevent musculoskeletal disorders. Participants will be assessed primarily for acceptability, suitability, feasibility, and fidelity, and secondarily for the occurrence of musculoskeletal complaint and the number of days from randomization on which this musculoskeletal complaint occurred, type of delivery and costs. Then, participants will be randomized into two groups: the usual care group, which will receive an educational booklet with information about the usual care during pregnancy, and the Pilates group, which will receive the same educational booklet and will participate in a specific Pilates exercise program for the gestational period, twice a week, throughout the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women of usual risk in the 12th gestational week (gestational age determined by the date of the last menstruation or by the ultrasound examination)
* with medical clearance to practice physical activity

Exclusion Criteria:

* practice of other physical activity during pregnancy
* any medical contraindications, such as diabetes and hypertension

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability measured using a 11-point numerical scale (0 = completely dissatisfied with the treatment results; 10 = completely satisfied with the treatment results) | 24th gestational week
  The participant's perception of the treatment result being satisfactory
Acceptability measured using a 11-point numerical scale (0 = completely dissatisfied with the treatment results; 10 = completely satisfied with the treatment results) | 36th gestational week
  The participant's perception of the treatment result being satisfactory
Acceptability measured using a 11-point numerical scale (0 = completely dissatisfied with the treatment results; 10 = completely satisfied with the treatment results) | From 7 to 15 days after delivery
  The participant's perception of the treatment result being satisfactory
Suitability measured using 2 questions (one about the need of tailored exercises for the gestational needs and the other about the need of some adaptation during the execution of the exercises) | 24th gestational week
  Assesses whether the exercise program is suitable for the target audience or needs some adaptation
Suitability measured using 2 questions (one about the need of tailored exercises for the gestational needs and the other about the need of some adaptation during the execution of the exercises) | 36th gestational week
  Assesses whether the exercise program is suitable for the target audience or needs some adaptation
Suitability measured using 2 questions (one about the need of tailored exercises for the gestational needs and the other about the need of some adaptation during the execution of the exercises) | From 7 to 15 days after delivery
  Assesses whether the exercise program is suitable for the target audience or needs some adaptation
Viability measured using a form developed for this study and filled by the physical therapist responsible for the treatment | 24th gestational week
  Assesses recruitment, retention, and participation rates, whether participants reached the end of the treatment program and, if not, why they dropped out
Viability measured using a form developed for this study and filled by the physical therapist responsible for the treatment | 36th gestational week
  Assesses recruitment, retention, and participation rates, whether participants reached the end of the treatment program and, if not, why they dropped out
Viability measured using a form developed for this study and filled by the physical therapist responsible for the treatment | From 7 to 15 days after delivery
  Assesses recruitment, retention, and participation rates, whether participants reached the end of the treatment program and, if not, why they dropped out
Fidelity measured using an exercise checklist (list of all exercises that can be performed including the level of difficulty) | 24th gestational week
  Assesses the level of difficulty of the selected exercises
Fidelity measured using an exercise checklist (list of all exercises that can be performed including the level of difficulty) | 36th gestational week
  Assesses the level of difficulty of the selected exercises
Fidelity measured using an exercise checklist (list of all exercises that can be performed including the level of difficulty) | From 7 to 15 days after delivery
  Assesses the level of difficulty of the selected exercises

SECONDARY OUTCOMES:
Occurrence of musculoskeletal complaint | 24th gestational week, 36th gestational week, and from seven to 15 days after delivery
Number of days from randomization on which the musculoskeletal complaint occurred | 24th gestational week, 36th gestational week, and from seven to 15 days after delivery
Delivery mode (normal or caesarean section) | From 7 to 15 days after delivery
Apgar score (0 to 10) | From 7 to 15 days after delivery
  Reported at 1 minute and 5 minutes after birth, and at 5-minute intervals thereafter until 20 minutes for infants with a score less than 7
Baby's birth weight | From 7 to 15 days after delivery
Kinesiophobia measured using the Tampa Scale of Kinesiophobia in the occurrence of musculoskeletal complaint | 24th gestational week, 36th gestational week, and from 7 to 15 days after delivery
  The total score ranges from 17 to 68 points, and the higher the score, the greater the degree of kinesiophobia.
Disability measured using the Patient Specific Functional Scale in the occurrence of musculoskeletal complaint | 24th gestational week, 36th gestational week, and from 7 to 15 days after delivery
  11-point numerical scale (0 = unable to perform the activity; 10 = able to perform the activity at the same level as before the injury or problem)
Pain measured using the Pain Numerical Rating Scale in the occurrence of musculoskeletal complaint | 24th gestational week, 36th gestational week, and from 7 to 15 days after delivery
  11-point numerical scale (0 = no pain; 10 = the worst possible pain)
Costs (healthcare costs, patient and family costs, and lost productivity costs) measured using a questionnaire specially developed for this study | Baseline, 24th gestational week, 36th gestational week, and from 7 to 15 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Cristina MN Cabral, PhD, Principal Investigator — Universidade Cidade de São Paulo

IPD SHARING:
Plan to Share IPD: Undecided